CLINICAL TRIAL: NCT00158977
Title: CONTAK RENEWAL 3 AVT Study
Brief Title: CONTAK RENEWAL 3 AVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0008
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: heart failure; atrial fibrillation; cardiac resynchronization therapy defibrillator
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

INTERVENTIONS:
Device: CONTAK RENEWAL 3 AVT — CONTAK RENEWAL 3 AVT

SUMMARY:
The RENEWAL 3 AVT device is designed to treat patients suffering from HF, with a history of or at risk of developing atrial and ventricular arrhythmias

DETAILED DESCRIPTION:
A clinical evaluation to:

* Confirm that there are no adverse interactions when Ventricular Tachyarrhythmia (ICD), Heart Failure (HF) and Atrial Tachyarrhythmia (AT) therapies are combined
* Confirm Cardiac Resynchronization Therapy (CRT) and Ventricular Tachyarrhythmia (ICD) therapy is delivered in the presence of atrial therapies
* Demonstrate the safety and effectiveness of atrial therapies in a heart failure population

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria should be given consideration for inclusion in the clinical investigation:

* Meet all device indications and contraindications
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigational center and at the intervals defined by this protocol
* Prescribed to stable optimal pharmacologic therapy for heart failure
* Creatinine < 2.5 mg/dL obtained no more than two weeks prior to enrollment
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Geographically stable residents who are available for follow-up
* Able to provide documented evidence of one or more episodes of AF/AT within 12 months of implantation

NOTE: Guidant recommends anticoagulation therapy per physician discretion.

Exclusion Criteria:

Patients who will be excluded from the investigation are those who meet any one of the following criteria:

* Have a preexisting non-Guidant left ventricular lead
* Have a preexisting unipolar pacemaker that will not be explanted/abandoned
* Documented life expectancy of less than six months or expected to undergo heart transplant within the next six months
* Have an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) within 180 days prior to enrollment
* Have a known hypersensitivity to a 0.7 mg dose of dexamethasone acetate
* Have surgically uncorrected primary valvular heart disease
* Currently requiring hemo-dialysis
* Have had a myocardial infarct, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the preceding 30 days prior to enrollment
* Have hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis)
* Have a mechanical tricuspid heart valve
* Enrolled in any concurrent study, without Guidant written approval, that may confound the results of this study
* A Cerebral Vascular Event/ Transient Ischemic Attack within 12 months of implantation
* During the four weeks prior to implantation, a patient experiences an episode of AF ³ 48 hours in duration and was not anticoagulated at an adequate therapeutic level for the 4 weeks prior to enrollment with an INR = 2.0-3.0 at enrollment
* Women who are pregnant or plan to become pregnant

Note: Women of childbearing potential must have a negative pregnancy test within 7 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-11; Primary Completion 2004-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint: To show that the RENEWAL 3 AVT system functions safely at 3 months | 3 months
Effectiveness Endpoint: To demonstrate the effective termination of induced episodes of atrial fibrillation by cardioversion | 3 months
Effectiveness Endpoint: To correctly detect and classify atrial arrhythmias (AF and/or SVT) from all other rhythms | 3 months

SECONDARY OUTCOMES:
Safety Endpoint: Ventricular Fibrillation (VF) Detection Time | 3 months
Safety Endpoint: Percent BiV Pacing | 3 months
Safety Endpoint: EASYTRAK 2 Lead Complication-Free Rate | 3 months
Safety Endpoint: Rate of Inappropriate Response to BiV Trigger Feature | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple locations in the US, Saint Paul, Minnesota, United States

REFERENCES:
- [Result] Saxon LA, Greenfield RA, Crandall BG, Nydegger CC, Orlov M, VAN Genderen R. Results of the multicenter RENEWAL 3 AVT clinical study of cardiac resynchronization defibrillator therapy in patients with paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2006 May;17(5):520-5. doi: 10.1111/j.1540-8167.2006.00440.x. PMID 16684026